CLINICAL TRIAL: NCT05499273
Title: Pediatric Neck Rescue: Randomized Comparison of Two Emergency Approaches to the Trachea in an Advanced Simulated Rabbit Model
Brief Title: Pediatric Neck Rescue Access Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Gaslini Children's Hospital (Other)
Responsible Party: Principal Investigator, Thomas Riva, PD Dr. med., Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Riva-Ulmer2022
Record Dates: First submitted 2022-06-24; First posted 2022-08-12 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Tracheostomy Complication; Anesthesia
Keywords: pediatric airway; tracheotomy; eFONA; CICO

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scalpel-bougie tracheostomy (SBT) (Active Comparator): SBT technique described in Interventions
  Interventions: Procedure: scalpel-bougie tracheostomy; Procedure: rapid sequence tracheotomy
- rapid sequence tracheotomy (RST (Active Comparator): RST technique described in Interventions
  Interventions: Procedure: scalpel-bougie tracheostomy; Procedure: rapid sequence tracheotomy

INTERVENTIONS:
Procedure: scalpel-bougie tracheostomy — 1. The assistant places themselves with two preparation clamps at the head end of the table and assists with each hand placed lateral to the neck, so that the operating field is freely accessible. After the trachea or cricoid is palpated, a long median longitudinal skin incision of 2-3 cm is made from the cricoid caudally
  2. The assistant uses straight clamps to pull the two edges of the skin incision apart dorso-laterally. In the event of major bleeding this maneuver should allow the blood to drain off dorsally and the view of the anatomical structures should be less impaired.
  3. Layer by layer of the anatomical structures are cut through with the scalpel and tightened with the clamps accordingly.
  4. Using a longitudinal incision, two to three tracheal rings are cut through distally to the cricoid
  5. An 8 FR Frova catheter is inserted through the orifice into trachea.
  6. A tracheal tube (ID 3.0 mm) is inserted over the Frova catheter to secure the airway permanently.
  Other Names: SBT
Procedure: rapid sequence tracheotomy — 1. Orientational palpation and vertical midline skin incision followed by separation of the strap muscles
  2. Exposure of the trachea and cricoid followed by anterior luxation of the trachea with a Backhaus towel clamp
  3. Perform a vertical puncture with a tip scissors between the cricoid and 1st tracheal ring followed by a vertical incision of no more than 2 rings in length.
  4. A tracheal tube (inner diameter 3.0 mm, cuffed) is inserted to secure the airway permanently.
  Other Names: RST

SUMMARY:
Two recent studies explored the emergency tracheotomy technique and the scalpel-bougie-tracheostomy technique as a neck rescue access for newborns and infants on a rabbit cadaver. Both studies lacked a key feature of real surgical access - bleeding during a true emergency. The study's objective was to comparatively assess the two techniques in a simulated environment with simulated bleeding and decreasing vital signs from the monitor like in real emergencies.

DETAILED DESCRIPTION:
With ethical committee's approval the investigarors recruited for this cross-over trial pediatric anesthesiologists and intensivists. Emergency tracheotomy consists of four steps: vertical skin incision, strap muscles separation (2 Backhaus clamps), anterior luxation of the trachea with a 3rd clamp, and vertical puncture with tip-scissors of no more than 2 tracheal rings to insert the tube. The scalpel-bougie-tracheostomy involves separation of neck tissues to expose the trachea and tracheal incision both with a scalpel to insert the bougie to facilitate tracheal intubation. Participants were randomized to start either with emergency tracheotomy or scalpel-bougie-tracheostomy. They watched an instructional video and had four practicing attempts, followed by a fifth attempt which was assessed. Afterward, they crossed over to the other technique.

ELIGIBILITY:
Inclusion Criteria:

* board certified pediatric anesthesiologists or pediatric intensive care doctor
* informed consent signed

Exclusion Criteria:

* none

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Performance Time | 2 min
  performance time between the rapid sequence tracheotomy technique and the scalpel-bougie tracheostomy technique.

SECONDARY OUTCOMES:
rate of cricoid injuries | 2 min
  rate of cricoid cartilage injuries during procedure, that would preclude ventilation measured in %
Succes rate | 2 min
  succes rate in %
rate of thyroid injuries | 2 min
  rate of thyroid cartilage injuries during the procedure that would preclude ventilation, measured in %
number of tracheal ring damaged | 2 min
  number of damaged tracheal rings and perforation of the posterior tracheal wall during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riva, MD, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Riva T, Goerge S, Fuchs A, Greif R, Huber M, Lusardi AC, Riedel T, Ulmer FF, Disma N. Emergency front-of-neck access in infants: A pragmatic crossover randomized control trial comparing two approaches on a simulated rabbit model. Paediatr Anaesth. 2024 Mar;34(3):225-234. doi: 10.1111/pan.14796. Epub 2023 Nov 10. PMID 37950428